CLINICAL TRIAL: NCT05537649
Title: Glycemic Responses of an Innovative Oat Porridge
Acronym: GREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S64889
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Postprandial Glycemic Responses
Keywords: enzymatic starch modification; postprandial glycemic responses

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oatmeal porridge (Active Comparator): Cold-stored oatmeal porridge (38 g oats) and stored for 24 h at 4 degrees Celsius
  Interventions: Dietary Supplement: Oatmeal porridge
- Oatmeal porridge treated with amylomaltase (Active Comparator): Cold-stored oatmeal porridge (38 g oats) treated with 30 enzyme units/g oats of amylomaltase and stored for 24 h at 4 degrees Celsius
  Interventions: Dietary Supplement: Oatmeal porridge

INTERVENTIONS:
Dietary Supplement: Oatmeal porridge — Investigation of the impact of enzymatic modification of the molecular structure of starch by amylomaltase on the postprandial glycemic responses of an oatmeal porridge.

SUMMARY:
The aim of this study is to investigate whether enzymatic modification of starch in a food product using amylomaltase induces a lower glycemic response in healthy subjects compared to its unmodified counterpart.

DETAILED DESCRIPTION:
A single-blind, randomized, cross-over study design will be applied. During each of the two study visits, healthy participants will consume an oatmeal porridge. One porridge will be treated will amylomaltase to modify the molecular structure of starch while the other porridge will serve as a control (unmodified counterpart). Blood glucose measurements will be taken postprandially at regular time points.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) range 18.5 - 25.0 kg/m2 at screening visit
* Fasting whole blood glucose values < 6.3 mmol/L
* Regular diet with 3 meals a day (at least 5 times a week)
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigators on the basis of medical history
* Willingness to maintain habitual diet, physical activity pattern, and body weight throughout the trial and refrain from smoking for 12 h prior to each visit
* Willingness to abstain from alcohol consumption and to avoid vigorous physical activity for 24 h prior to study visits.
* Adequate level of understanding spoken and written English
* Willingness to provide informed consent to participate in the study

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Recent participation in any clinical trial (< 90 days)
* Pregnant or lactating in the period of the study
* Known history of AIDS, hepatitis, diabetes mellitus (Type I and II), cardiovascular disease, any pathology (or recent surgical event) of the gastrointestinal system or any current metabolic or endocrine disease
* Alcohol consumption of > 14 standard drinks for women and > 21 standard drinks for men per week
* Celiac disease or gluten intolerance
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids the last 4 weeks before the screening visit
* Use of antibiotics during the last three months
* Reported slimming or medically prescribed diet
* Unwillingness or inability to comply with the experimental procedures and to follow the safety guidelines

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Glucose response | up to 3 hours
  incremental area under the curve of blood glucose after oat porridge consumption

SECONDARY OUTCOMES:
Glucose response | up to 3 hours
  peak rise of the blood glucose after oat porridge consumption

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Vlaams-Brabant, Belgium